CLINICAL TRIAL: NCT00111501
Title: LGBT Internet Based Smoking Treatment
Brief Title: LGBT Internet Based Smoking Treatment - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-15791-1; R01DA015791 (NIH); R01-15791-1
Record Dates: First submitted 2005-05-20; First posted 2005-05-23 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Tobacco Use Disorder
Keywords: smoking; tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted Internet Intervention (Experimental): Web-based self help intervention developed to include specific cultural tailoring relevant to the LGBT community
  Interventions: Behavioral: Tobacco Use Disorder
- Standard Intervention (Active Comparator): Standard self-help internet-based intervention with no LGBT relevant information included
  Interventions: Behavioral: Standard Web-based intervention

INTERVENTIONS:
Behavioral: Tobacco Use Disorder — Web-based psychoeducational intervention culturally-tailored to the LGBT community including a social support component
  Arms: Targeted Internet Intervention
Behavioral: Standard Web-based intervention — General psychoeducational Web-based smoking cessation intervention
  Arms: Standard Intervention

SUMMARY:
The overall goals of this line of research are to develop and evaluate innovative treatments for lesbian, gay, bisexual, and transgender (LGBT) cigarette smokers and to understand the processes related to smoking and relapse in this previously unstudied population of smokers. In this study, participants are randomly assigned to one of two Internet-based smoking cessation treatments: 1) a self-help intervention tailored LGBT smokers plus social support plus email-based counseling, or 2) a standard self-help condition alone, similar to other general smoking cessation treatments. Before starting the program, participants will complete measures of smoking, nicotine dependence, depression diagnosis, demographics, mood, motivation to change, and alcohol use. Smoking status will be determined at 1, 3, 6, and 12 months following the start of treatment. Data will be analyzed to compare the quit rates of the two Internet-based treatment groups. Also, we will complete exploratory analyses to determine those variables that best predict quitting for LGBT smokers.

ELIGIBILITY:
Must identify as a lesbian, gay male, bisexual male or female or a transgender individual. Must smoke most days during the preceding month. Must have a valid email address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 792 (Actual)
Dates: Start 2002-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
point-prevalence abstinence from tobacco use | 7-day
  Self-report of smoking status during the past seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Humfleet, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Medical Cen, San Francisco, California, United States